CLINICAL TRIAL: NCT06574958
Title: Professor of Medicine Second Hospital of Shandong University
Brief Title: Clinical Study of CD38\CS1 Chimeric Antigen Receptor T Cells in the Treatment of Refractory/Recurrent Multiple Myeloma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Linlin Cui, professor of medicine, The Second Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 CD38/CS1 T cell of MM
Record Dates: First submitted 2024-08-13; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: ORR,OS,PFS

STUDY DESIGN:
Intervention Model Description: 10
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- refractory or relapsed MM (Experimental)
  Interventions: Biological: CD38/CS1 injection

INTERVENTIONS:
Biological: CD38/CS1 injection — Dosage form and specification: injection, 40mL/ dose, according to the number of positive cells 1×106/kg Properties: Colorless or slightly light white clear liquid Prescription composition: CD38/CS1 CAR T cells, 2.5% human blood albumin, 0.9% sodium chloride injection.
  Administration mode: intravenous injection Storage condition: 2-8℃ for 8h Mechanism of action :38WP as a dual-target CAR T cell therapy, compared with single-target CAR T cell therapy, its advantage is that it can reduce antigen escape of tumor cells.

SUMMARY:
The investigators developed a dual-target CAR-T targeting CD38 and CS1. Previous experimental results showed that the investigators double-target CAR-T not only had a good killing effect on CD38/CS1 double-positive tumor cells, but also had a high killing rate on CD38 or CS1 single-positive tumor cells. The investigators further study also found that the killing rate of the investigators dual-target CAR-T after mixing CD38 and CS1 monoyang tumor cells was over 80%. The advantage of the investigators dual-target CAR-T product is that the killing effect on single-yang, double-yang and single-yang mixed tumors is stable, and the killing rate is above 80% (see Figure 1). It has a wide killing range and can effectively reduce the phenomenon of tumor immune escape. Therefore, the investigators dual CAR products have good advantages and development potential.

ELIGIBILITY:
Inclusion Criteria:1. Relapsed, refractory, drug-resistant MM. 2. MM patients who have not achieved CR in 4 cycles of standard treatment. 3. Age over 15 and under 75. 4. KPS≥50 or ECOG score ≤2 points and expected survival greater than 3 months. 5. No systemic therapy (except systemic immune checkpoint suppression or activation therapy) for at least 2 weeks or at least 5 drug half-lives (whichever is shorter) prior to apheresis. 6. The absolute number of neutrophils was > 1.0x109 /L. 7. Absolute number of platelets > 50x109 /L. 8. Absolute number of lymphocytes ≥ 0.15x109 /L. 9. ALT/AST < 3 times the normal value. 10. Total bilirubin < 1.5mg/dl. 11. Creatinine < 2.5mg/dl, or creatinine clearance ≥60 mL/min/1.73 m2. 12. Cardiac ejection fraction ≥ 45%, echocardiography (ECHO) showed no pericardial effusion, electrocardiogram (ECG) was normal 13. Blood oxygen saturation ≥92% under normal conditions. 14. Women of childbearing age who had a negative urine pregnancy test before the start of dosing and consented to effective contraceptive use during the trial period until the last follow-up visit. 15. Volunteer to participate in this experiment and sign the informed consent.

-

Exclusion Criteria:1. Patients with expected survival of less than 3 months. 2. Patients whose disease progression was so rapid that a complete treatment cycle could not be ensured according to the investigator at the time of enrollment. 3. Patients with primary tumors other than melanoma skin cancer (e.g. cervical cancer, bladder cancer, breast cancer) (unless cured for more than 3 years). 4. Patients with infections including fungal, bacterial, viral or other uncontrolled infections or those requiring level 4 isolation. 5. Patients who test positive for HIV, HBV and HCV. 6. Patients with central nervous system diseases including stroke, epilepsy, dementia or autoimmune central nervous system diseases. 7. Patients with myocardial infection, cardiac angiography or stent, active angina pectoris or other significant clinical symptoms, or with cardiogenic asthma or cardiovascular plasma cell infiltration in the 12 months prior to enrollment. 8. People who are receiving anticoagulant therapy or have severe coagulation disorders. 9. According to the judgment of the researcher, the drug treatment that the patient is receiving will affect the safety and effectiveness study of this project. 10. Patients with allergy or history of allergy to the biologics used in this project. 11. Pregnant or lactating women. 12. Systematic use of systemic or systemic steroid drugs within 2 weeks prior to treatment (except those who have recently or currently used inhaled steroids). 13. The efficiency of T cell transduction by replication-deficient lentivirus is less than 30%, or the amplification ability is insufficient (times) in response to CD3 / CD28 co-stimulatory signals. 14. Patients with other uncontrolled diseases deemed unsuitable by the researchers. 15. Any situation that the investigator believes may increase the risk to the subject or interfere with the test results. 16. Patients who are also participating in other clinical studies.

-

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
ORR | one year
  sCR、CR、VGPR、PR

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shandong University, Shandong, Shandong, China

IPD SHARING:
Plan to Share IPD: No